CLINICAL TRIAL: NCT04504721
Title: Effects of Blue-enriched White Light Therapy on Sleep Quality, Depression, Psychomotor Vigilance, and Symptom Severity in Patients with Fibromyalgia
Brief Title: Effects of Blue-enriched White Light Therapy in Patients with Fibromyalgia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Pei-Shan, Tsai, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: N202003152
Record Dates: First submitted 2020-08-06; First posted 2020-08-07 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-11

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Light therapy; Sleep quality; Depression
MeSH Terms: conditions — Fibromyalgia; Sleep Initiation and Maintenance Disorders; Depression | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Light therapy group (Experimental): The intervention will take 8 weeks with 30 minutes exposure at awakening to blue-enriched white light.
  Interventions: Other: light therapy
- Waiting list group (No Intervention): Participants who are randomly assigned into the waiting list group will be told that they are on a waiting list to be enrolled in the study. Participants will be provided with light therapy after the first posttest outcome assessments are completed.

INTERVENTIONS:
Other: light therapy — The intervention will take 8 weeks with 30 minutes exposure at awakening to blue-enriched white light.
  Arms: Light therapy group

SUMMARY:
Fibromyalgia is a chronic condition with an unclear etiology. The syndrome includes symptoms such as chronic musculoskeletal pain, cognitive dysfunctions, fatigue, sleep disorders, and circadian rhythm disturbances. Fibromyalgia-related pain is associated with a substantial socioeconomic burden including greater health care costs and productivity loss from work. Light therapy can improve sleep quality and sleep architecture, advance sleep phases and reduce pain sensitivity and that the effect of light therapy on mood and cognitive function have been widely supported.This randomized controlled study aims to examine the effects of light therapy on sleep quality, depressive symptoms, psychomotor vigilance performance, and overall symptom severity in patients with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is a central sensitivity syndrome characterized by chronic widespread pain, cognitive dysfunctions, fatigue, sleep disorders, and circadian dysregulation. Light therapy can improve sleep quality and sleep architecture, advance sleep phases and reduce pain sensitivity and that the effect of light therapy on mood and cognitive function have been widely supported, research into the effect of light therapy for patients with fibromyalgia who often suffer from sleep and mood disturbance, pain, and cognitive impairments is of both research interest and therapeutic implications. This study will use a randomized, parallel group, assessor-blind, waiting-list controlled trial design. The primary outcome is symptom severity. The secondary outcomes include: sleep quality; depressive symptoms; psychomotor vigilance and attention; and sleep phase changes. The intervention will take 8 weeks with 30 minutes exposure at awakening to blue-enriched white light. A total of 80 participants, aged 20 to 64, with a diagnosis of fibromyalgia will be enrolled and randomly assigned into one of the two parallel groups: an intervention and a waiting list group. For the intervention group, outcomes will be assessed at baseline, immediately after, and 2 months after the 8-week intervention period. For the waiting list group, outcomes will be assessed at baseline, immediately after the 8-week waiting period, and 2 months after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be aged from 20 to 64 years old.
2. Participants must read and understand Chinese language.
3. Participants must be outpatients.
4. Participants must have a confirmed diagnosis of fibromyalgia according to the 2016 American College of Rheumatology diagnostic criteria.

Exclusion Criteria:

1. Subjects who are admitted to the hospital.
2. Subjects who have other significant chronic disease, past or present psychosis, or bipolar disorder.
3. Subjects who have ophthalmic pathology (cataract, macular degeneration, glaucoma, retinitis pigmentosa), eye surgery, diseases affecting the retina (retinopathy, diabetes, herpes, etc.), color blind, or taking photosensitizing medications.
4. Subjects who are taking opiates or benzodiazepines.
5. Subjects who work night shifts, or travel across more than two time zones in the month prior to enrolling in the study.
6. Subjects who are pregnant.
7. Subjects who have used light treatment in the last 6 months.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire-Revised Version | Baseline
  Fibromyalgia symptom severity will be measured using the Fibromyalgia Impact Questionnaire-Revised Version (FIQR) .The FIQR contains a total of 21 individual questions in three domains: function, impact and symptom domains. All questions are based on an 11-point numeric rating scale of 0 to 10, with '0' representing 'no difficulty' and '10' representing 'worst'.
Fibromyalgia Impact Questionnaire-Revised Version | Immediately after the 8-week intervention period
  Fibromyalgia symptom severity will be measured using the Fibromyalgia Impact Questionnaire-Revised Version (FIQR) .The FIQR contains a total of 21 individual questions in three domains: function, impact and symptom domains. All questions are based on an 11-point numeric rating scale of 0 to 10, with '0' representing 'no difficulty' and '10' representing 'worst'.
Fibromyalgia Impact Questionnaire-Revised Version | 2 months after the 8-week intervention period
  Fibromyalgia symptom severity will be measured using the Fibromyalgia Impact Questionnaire-Revised Version (FIQR) .The FIQR contains a total of 21 individual questions in three domains: function, impact and symptom domains. All questions are based on an 11-point numeric rating scale of 0 to 10, with '0' representing 'no difficulty' and '10' representing 'worst'.

SECONDARY OUTCOMES:
Sleep quality | Baseline
  The Pittsburgh Sleep Quality Index (PSQI) is a self-administered questionnaire that assesses sleep quality over a 1-month time interval. The seven components include subjective sleep quality, sleep latency, total sleep time, habitual sleep efficiency, sleep disorders, use of sleep medications, and daytime dysfunction. All questions are scored on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where higher scores denote a poorer sleep quality.
Sleep quality | Immediately after the 8-week intervention period
  The Pittsburgh Sleep Quality Index (PSQI) is a self-administered questionnaire that assesses sleep quality over a 1-month time interval. The seven components include subjective sleep quality, sleep latency, total sleep time, habitual sleep efficiency, sleep disorders, use of sleep medications, and daytime dysfunction. All questions are scored on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where higher scores denote a poorer sleep quality.
Sleep quality | 2 months after the 8-week intervention period
  The Pittsburgh Sleep Quality Index (PSQI) is a self-administered questionnaire that assesses sleep quality over a 1-month time interval. The seven components include subjective sleep quality, sleep latency, total sleep time, habitual sleep efficiency, sleep disorders, use of sleep medications, and daytime dysfunction. All questions are scored on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where higher scores denote a poorer sleep quality.
Depressive symptoms | Baseline
  The Beck Depression Inventory Version 2 (BDI-II) is a self-report 21-item questionnaire in which responses are rated on a 0 to 3 interval scale, with a higher score denoting mire frequent symptoms. The possible score of BDI-II ranges from 0 to 63, with higher scores representing more sever ratings of depression.
Depressive symptoms | Immediately after the 8-week intervention period
  The Beck Depression Inventory Version 2 (BDI-II) is a self-report 21-item questionnaire in which responses are rated on a 0 to 3 interval scale, with a higher score denoting mire frequent symptoms. The possible score of BDI-II ranges from 0 to 63, with higher scores representing more sever ratings of depression.
Depressive symptoms | 2 months after the 8-week intervention period
  The Beck Depression Inventory Version 2 (BDI-II) is a self-report 21-item questionnaire in which responses are rated on a 0 to 3 interval scale, with a higher score denoting mire frequent symptoms. The possible score of BDI-II ranges from 0 to 63, with higher scores representing more sever ratings of depression.
Psychomotor vigilance and attention | Baseline
  Psychomotor vigilance and attention will be measured using the Psychomotor Vigilance Task (PVT). The visual stimulus and performance feedback are presented on the device.
Psychomotor vigilance and attention | Immediately after the 8-week intervention period
  Psychomotor vigilance and attention will be measured using the Psychomotor Vigilance Task (PVT). The visual stimulus and performance feedback are presented on the device.
Psychomotor vigilance and attention | 2 months after the 8-week intervention period
  Psychomotor vigilance and attention will be measured using the Psychomotor Vigilance Task (PVT). The visual stimulus and performance feedback are presented on the device.
Sleep phase assessment | Baseline
  The Morningness-Eveningness Questionnaire (MEQ) is used to estimate phase preferences in circadian rhythms based on participants' self-descriptions. timing. Questions evaluate the time that individuals get up and go to bed, self-reported preferred times for physical and mental activity, and also the individual's subjective alertness. MEQ scores can range from 16 to 86, with lower scores indicating eveningness or later circadian timing, and higher scores indicating morningness or earlier circadian timing.
Sleep phase assessment | Immediately after the 8-week intervention period
  The Morningness-Eveningness Questionnaire (MEQ) is used to estimate phase preferences in circadian rhythms based on participants' self-descriptions. timing. Questions evaluate the time that individuals get up and go to bed, self-reported preferred times for physical and mental activity, and also the individual's subjective alertness. MEQ scores can range from 16 to 86, with lower scores indicating eveningness or later circadian timing, and higher scores indicating morningness or earlier circadian timing.
Sleep phase assessment | 2 months after the 8-week intervention period
  The Morningness-Eveningness Questionnaire (MEQ) is used to estimate phase preferences in circadian rhythms based on participants' self-descriptions. timing. Questions evaluate the time that individuals get up and go to bed, self-reported preferred times for physical and mental activity, and also the individual's subjective alertness. MEQ scores can range from 16 to 86, with lower scores indicating eveningness or later circadian timing, and higher scores indicating morningness or earlier circadian timing.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Shan Tsai, PhD, Study Chair — Taipei Medical University
Locations (1):
- Bio-Behavior Research Laboratory, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No